CLINICAL TRIAL: NCT01399801
Title: Optimizing the Left Ventricular Contractility in Cardiac Resynchronization Therapy Using a Doppler Wire
Brief Title: Optimizing Left Ventricular Lead To Improve Cardiac Output
Acronym: CARE/VOLCANO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann Marie Chikowski (Other)
Collaborators: Main Line Health (Other)
Responsible Party: Sponsor-Investigator, Ann Marie Chikowski, Division Manager Cardiology Research, Main Line Health
Organization: Main Line Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F/N-R09-284IL
Record Dates: First submitted 2011-06-16; First posted 2011-07-22 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Ischemic Congestive Cardiomyopathy; Dilated Cardiomyopathy; Congestive Heart Failure
Keywords: Cardiac Resynchronization Therapy; medically refractory heart failure patients
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hemodynamicaly guided LV lead placement (Experimental): optimized left ventricular lead placement
  Interventions: Procedure: Doppler flow measurement
- Standard lead placement (Active Comparator): Standard LV lead placement with no measurements to guide LV lead placement
  Interventions: Procedure: standard implantation of the LV lead

INTERVENTIONS:
Procedure: Doppler flow measurement — use of doppler wire to measure change in flow that corresponds to changes in stroke volume to guide LV lead placement
  Arms: hemodynamicaly guided LV lead placement
Procedure: standard implantation of the LV lead — Standard implantation of the LV lead with measurements of flow
  Arms: Standard lead placement

SUMMARY:
The purpose of this study is to determine if optimal lead placement, guided by the largest improvement in aortic flow measured by Doppler will:

1. Improve the way the heart's left ventricle functions
2. Decrease the number of hospital admissions for heart failure related symptoms
3. Reduces uncoordinated heart contractions
4. Improve quality of life as measured by the Minnesota Living with Heart Failure Questionaire and NYHA Class assessed after six months

DETAILED DESCRIPTION:
The hypothesis of this study determines if response to CRT therapy could be improved by optimizing LV lead position at the time of the left ventricular pacing lead implantation. This optimization (using a Doppler wire) would alter the left ventricular activation pattern and contraction mechanics. This increase in contractility may improve the likelihood of mid/long term response to therapy. This study will compare 6-month response to CRT (left ventricular ejection fraction, decrease in left ventricular end systolic and end diastolic dimensions and volumes) in heart failure patients.

The secondary objective will be to:

1. To determine if optimal lead placement, guided by the largest improvement in stroke volume, results in a greater 6-month improvement in clinical QOL and NYHA class.
2. Acutely compare and/or correlate intra-operative A-V and V-V timing optimization via invasive pressure volume data to post-operative echo optimization of these same parameters.
3. Acutely contrast changes in stroke volume during pacing from several different left ventricular lead locations.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for CRT-P or CRT-D
* QRS Duration>=120 MSEC
* Left Ventricular Ejection fraction<=35%
* NYHA Class III-IV
* History of Cardiomyopathy, least one month post MI, or at least six months old in case of non-ischemic cardiomyopathy
* At least 18 years of afe

Exclusion Criteria:

* Previous implanted CRT-P/CRT-D
* woman who are pregnant
* Psychological or emotional problems

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2014-09-25 (Actual); Study Completion 2014-09-25 (Actual)

PRIMARY OUTCOMES:
Change in Left Ventricular End Systolic Volume (LVESV) using the difference from baseline to six months | Six months
  Comparison of clinical and functional outcomes of stroke volume optimized lead placement to standard lateral lead placement.

SECONDARY OUTCOMES:
Change in End diastolic volume | Six months
  End diastolic volume should decrease over follow up time of six months as a result of left ventricular remodeling.
Change in ejection fraction | six months
  Increase in ejection fraction should happen as a result of remodeling and increased efficiency of the left ventricle
Increase in exercise capacity | six months
  Inrease in exercise capacity should be result of remodeled left ventricle and increased stroke volume and cardiac output
Decrease in heart failure related hospital admissions | six months
  number of hospitalizations for CHF should decrease during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Dusan Kocovic, MD, Principal Investigator — Lankenau Hospital
Locations (1):
- Lankenau Hosspital, Wynnewood, Pennsylvania, United States